CLINICAL TRIAL: NCT07000682
Title: Clinical Study on the Treatment of Refractory Moderate-to-Severe Active Systemic Sclerosis With UTAA91 Injection
Brief Title: The Clinical Study on the Treatment of SSc With UTAA91 Injection.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Qiubai Li, Director, Head of Department of Rheumatology and Immunology, Principal Investigator, Professor, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-010-9 (1)
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Systemic Sclerosis (SSc)
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: After signing the informed consent form, eligible subjects will be infused with UTAA91 injection. Blood samples will be collected from the subjects before and after the infusion for the evaluation of pharmacokinetics, pharmacodynamics, immunogenicity, safety, etc.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UTAA91 injection (Experimental)
  Interventions: Biological: UTAA91 injection

INTERVENTIONS:
Biological: UTAA91 injection — CAR-modified gamma delta T cells

SUMMARY:
This clinical trial is designed as a single-arm, open-label, single-center investigator-initiated early-phase study, with the primary objective of evaluating the safety of UTAA91 injection in subjects with refractory moderate-to-severe active systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years (inclusive of the boundary value), with no restriction on gender.

Expected survival time of ≥3 months. Refractory moderate - to - severe active systemic sclerosis that has failed standard treatment or lacks effective therapeutic options.

Meets the requirements for liver and kidney function, as well as cardiopulmonary function.

Free from severe psychiatric disorders. Able to understand the trial and has signed the informed consent form.

Exclusion Criteria:

* A history of malignant tumors other than relapsed/refractory autoimmune diseases (R/R AID) within 5 years prior to screening.

Positive results in virology/syphilis tests. Severe cardiac diseases or unstable systemic diseases. Presence of active or uncontrollable infections requiring systemic treatment, or evidence of central nervous system invasion.

Pregnant or breastfeeding women, female subjects planning to become pregnant within 2 years after cell infusion, or male subjects whose partners plan to become pregnant within 2 years after their cell infusion.

Subjects who have received CAR - T therapy or other gene - modified cell therapies prior to screening.

Subjects who participated in other clinical studies within 1 month prior to screening.

Other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | About 1 year
  The types, frequency, and severity of adverse events (AEs) and laboratory abnormalities (according to the Common Terminology Criteria for Adverse Events, NCI CTCAE 5.0).

SECONDARY OUTCOMES:
Cmax | About 1 year
  Maximum concentration of UTAA91 injection amplified in peripheral blood after administration of the drug
Tmax | About 1 year
  Time to reach maximum concentration in peripheral blood after administration of UTAA91 injection
Disease remission rate | About 3 months
  The disease remission/response/improvement rates at 28 days, 2 months, and 3 months after treatment with UTAA09 injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China